CLINICAL TRIAL: NCT05578885
Title: Dexamethasone Versus Fentanyl as an Adjuvant to Lidocaine in Bier Block for Patients Undergoing Hand Surgery
Brief Title: Duration of Analgesia in Bier Block for Patients Undergoing Hand Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michael Bishay Shehata Keroles (Other)
Responsible Party: Sponsor-Investigator, Michael Bishay Shehata Keroles, Resident doctor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IVRA
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Regional Anesthesia
Keywords: Dexamethasone; Intravenous regional anesthesia; Fentanyl; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Placebo Comparator): will receive Lidocaine
  Interventions: Procedure: Bier block
- Group B (Active Comparator): will receive Lidocaine Plus fentanyl
  Interventions: Procedure: Bier block
- Group C (Active Comparator): will receive lidocaine Plus dexamethasone
  Interventions: Procedure: Bier block

INTERVENTIONS:
Procedure: Bier block — patients in group a (n = 25) received 2% lidocaine3 mg/kg (maximum, 200 mg) for IVRA and 2 mL NaCl 0.9% IV , patients in group b (n = 25) received 2% lidocaine 3 mg/kg (maximum, 200 mg) plus 8 mg dexamethasone for IVRA and 2 mL NaCl 0.9% IV , and those in group c (n = 25) received 2% lidocaine 3 mg/kg (maximum, 200 mg) plus fentanyl IV

SUMMARY:
Intravenous regional anesthesia (Bier block) is widely used as an anesthetic technique for operations of short duration of the distal upper or lower extremities Today, IVRA is still popular in many countries being used in the emergency room, for outpatients and for high-risk patients with contraindications for general anesthesia.

DETAILED DESCRIPTION:
IVRA offers a favorable risk-benefit ratio, cost-effectiveness, sufficient muscle relaxation and a fast on- and offset. New upcoming methods for monitoring, specialized personnel and improved emergency equipment made IVRA even safer. Moreover, IVRA may be applied to treat complex regional pain syndromes. Prilocaine and lidocaine are considered as first-choice local anesthetics for IVRA. Also, various adjuvant drugs have been tested to augment the effect of IVRA, and to reduce post-deflation tourniquet pain. Since major adverse events are rare in IVRA, it is regarded as a very safe technique. Nevertheless, systemic neuro- and cardiotoxic side effects may be linked to an uncontrolled systemic flush-in of local anesthetics and must be avoided.

Dexamethasone decreases postoperative pain and prolongs the duration of local anaesthetic peripheral nerve blocks in studies including a limited number of patients .

Fentanyl is a powerful synthetic opioid that is similar to morphine but is 50 to 100 times more potent.fentanyl acts on opioid receptors. These receptors are G-protein-coupled receptors, which contain seven transmembrane portions, intracellular loops, extracellular loops, intracellular C-terminus, and extracellular N-terminus. The extracellular N-terminus is important in differentiating different types of binding substrates. When fentanyl binds, downstream signaling leads to the inhibitory effects, such as decreased cAMP production, decreased calcium ion influx, and increased potassium efflux. This inhibits the ascending pathways in the central nervous system to increase pain threshold by changing the perception of pain; this is mediated by decreasing propagation of nociceptive signals, resulting in analgesic effects

ELIGIBILITY:
Inclusion Criteria:

* ASA Grade 1 & 2

Exclusion Criteria:

Patient refusal ASA Grade 3 & 4 patients SEVERLY HYPOVOLEMIC STATE History of neurological. Reynauds disease, scleroderma, sickle cell anemia, myasthenia gravis, decompensated cardiac disease, diabetes mellitus, peptic ulcer, gastritis, and those with liver or renal insufficiency were excluded

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Compare duration of analgesia | one hour After procedure
  Change in the time of analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shehata, Resident, Principal Investigator — Assiut University; Eman Ismail, Professor, Study Director — Assiut University; Alaa Atia, Professor, Study Director — Assiut University
Locations (1):
- Faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No